CLINICAL TRIAL: NCT02561455
Title: A Phase 1/2 Open-label Rollover Study for Subjects Who Have Participated in an Astellas Sponsored ASP2215 Trial
Brief Title: Rollover Study for Subjects Who Have Participated in an Astellas Sponsored ASP2215 Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-0109
Expanded Access: NCT03070093 (Approved for marketing)
Record Dates: First submitted 2015-09-25; First posted 2015-09-28 (Estimated); Results first posted 2021-08-16 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumors; Acute Myeloid Leukemia
Keywords: Advanced solid tumors; Acute myeloid leukemia; gilteritinib; ASP2215
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Gilteritinib 40 mg (Experimental): Participants received gilteritinib 40 milligrams (mg) dose (one tablet of 40 mg) orally once a day in continuous 28-day cycles at least 2 hours after or 1 hour before food. Gilteritinib treatment continued until participants no longer received clinical benefit from therapy, or unacceptable toxicity occured, or met one of the treatment discontinuation criteria.
  Interventions: Drug: Gilteritinib
- Gilteritinib 80 mg (Experimental): Participants received gilteritinib 80 mg dose (two tablets of 40 mg) orally once a day in continuous 28-day cycles at least 2 hours after or 1 hour before food. Gilteritinib treatment continued until participants no longer received clinical benefit from therapy, or unacceptable toxicity occured, or met one of the treatment discontinuation criteria.
  Interventions: Drug: Gilteritinib
- Gilteritinib 120 mg (Experimental): Participants received gilteritinib 120 mg dose (three tablets of 40 mg) orally once a day in continuous 28-day cycles at least 2 hours after or 1 hour before food. Gilteritinib treatment continued until participants no longer received clinical benefit from therapy, or unacceptable toxicity occured, or met one of the treatment discontinuation criteria.
  Interventions: Drug: Gilteritinib
- Gilteritinib 200 mg (Experimental): Participants received gilteritinib 200 mg dose (five tablets of 40 mg) orally once a day in continuous 28-day cycles at least 2 hours after or 1 hour before food. Gilteritinib treatment continued until participants no longer received clinical benefit from therapy, or unacceptable toxicity occured, or met one of the treatment discontinuation criteria.
  Interventions: Drug: Gilteritinib

INTERVENTIONS:
Drug: Gilteritinib — oral tablet
  Other Names: ASP2215

SUMMARY:
The purpose of the study was to provide access to continued treatment for those who participated in other Astellas sponsored ASP2215 trials that completed the primary analysis and, had the potential to continue to derive clinical benefit from the treatment with ASP2215, and who did not meet any of the study discontinuation criteria in the present study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must currently be participating in an Astellas sponsored, single agent ASP2215 trial, receiving ASP2215 and have not met any discontinuation criteria of the parent study and can enroll into this rollover study without interruption of study drug, or with no more than 2 weeks interruption in study drug.
* Subject must be deriving benefit from continued treatment without any persistent intolerable toxicity from continued treatment of ASP2215.
* Female subject must either:

  * Be of non-childbearing potential: post-menopausal (defined as at least 1 year without any menses) prior to Screening, or documented surgically sterile or post-hysterectomy (at least 1 month prior to Screening)
  * Or, if of childbearing potential, Agree not to try to become pregnant during the study and for 180 days after the final study drug administration; And have a negative urine pregnancy test at Day 1; And, if heterosexually active, agree to consistently use two forms of highly effective birth control (at least one of which must be a barrier method) starting at Screening and throughout the study period and for 180 days after the final study drug administration.
* Female subject must agree not to breastfeed starting at Screening and throughout the study period, and for 60 days after the final study drug administration.
* Female subject must not donate ova starting at Screening and throughout the study period, and for 180 days after the final study drug administration.
* Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of two forms of birth control (at least one of which must be a barrier method) starting at Screening and continue throughout the study period, and for 120 days after the final study drug administration.
* Male subject must not donate sperm starting at Screening and throughout the study period and, for 120 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while on treatment.

Exclusion Criteria:

* Subject requires treatment with concomitant drugs that are strong inducers of cytochrome P450 (CYP)3A.
* Subject requires treatment with concomitant drugs that target serotonin 5-hydroxytryptamine receptor 1 (5HT1R) or 5-hydroxytryptamine receptor 2B (5HT2BR) or sigma nonspecific receptor with the exception of drugs that are considered absolutely essential for the care of the subject.
* Subject requires treatment with concomitant drugs that are strong inhibitors or inducers of P-glycoprotein (P-gp) with the exception of drugs that are considered absolutely essential for the care of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (7):
- United States (7):
  - Site US10005, Phoenix, Arizona
  - Site US10003, Baltimore, Maryland
  - Site US10006, New York, New York
  - Site US10007, New York, New York
  - Site US10001, Cleveland, Ohio
  - Site US10004, Hershey, Pennsylvania
  - Site US10008, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/patientStudySearch.aspx?RID=;;;2215-CL-0109

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from previosuly conducted ASP2215 trial were recruited to receive gilteritinib at a dose specified at the time of their end of study visit in the previous ASP2215 study.
Pre-assignment Details: Participants with Acute myeloid leukemia (AML) and advanced solid tumors who completed the protocol requirements of the previous ASP2215 trial (NCT02014558 and NCT02456883) were included in this study. 9 participants were screened.
Groups:
- Gilteritinib 40 mg: Participants received gilteritinib 40 milligrams (mg) dose (one tablet of 40 mg) orally once a day in continuous 28-day cycles at least 2 hours after or 1 hour before food. Gilteritinib treatment continued until participants no longer received clinical benefit from therapy, or unacceptable toxicity occurred, or met one of the treatment discontinuation criteria.
- Gilteritinib 80 mg: Participants received gilteritinib 80 mg dose (two tablets of 40 mg) orally once a day in continuous 28-day cycles at least 2 hours after or 1 hour before food. Gilteritinib treatment continued until participants no longer received clinical benefit from therapy, or unacceptable toxicity occurred, or met one of the treatment discontinuation criteria.
- Gilteritinib 120 mg: Participants received gilteritinib 120 mg dose (three tablets of 40 mg) orally once a day in continuous 28-day cycles at least 2 hours after or 1 hour before food. Gilteritinib treatment continued until participants no longer received clinical benefit from therapy, or unacceptable toxicity occurred, or met one of the treatment discontinuation criteria.
- Gilteritinib 200 mg: Participants received gilteritinib 200 mg dose (five tablets of 40 mg) orally once a day in continuous 28-day cycles at least 2 hours after or 1 hour before food. Gilteritinib treatment continued until participants no longer received clinical benefit from therapy, or unacceptable toxicity occurred, or met one of the treatment discontinuation criteria.
Period: Overall Study
Arm/Group | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg
Started | 2 | 3 | 3 | 1
Completed | 0 | 1 | 0 | 0
Not Completed | 2 | 2 | 3 | 1
Not completed — Participant Transitioned to Commercial Drug | 1 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Disease Progression | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population was the safety analysis set (SAF), which consisted of all participants who received at least 1 dose of study drug.
Groups:
- Gilteritinib 40 mg: Participants received gilteritinib 40 mg dose (one tablet of 40 mg) orally once a day in continuous 28-day cycles at least 2 hours after or 1 hour before food. Gilteritinib treatment continued until participants no longer received clinical benefit from therapy, or unacceptable toxicity occurred, or met one of the treatment discontinuation criteria.
- Total: Total of all reporting groups
Arm/Group | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Total
Number analyzed (Participants) | 2 | 3 | 3 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.5 (17.7) | 41 (17.5) | 55.7 (12.1) | 31.0 | 46.2 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 1 | 6
  Male | 0 | 2 | 1 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 2 | 2 | 3 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 3 | 3 | 1 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status was used to assess participants disease progression, and ability to carry out the daily living activities. Grade 0 = fully active, able to carry on all pre disease performance without restriction; Grade 1 = restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    Grade 0 | 1 | 2 | 0 | 1 | 4
    Grade 1 | 1 | 1 | 3 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: AE was defined as any untoward medical occurrence in a participant administered a study drug or has undergone study procedures and which did not necessarily have a causal relationship with this treatment. An abnormality identified during a medical test (e.g., laboratory parameter, vital sign, Electrocardiography (ECG) data, and physical exam) was defined as an AE only if the abnormality induces clinical signs or symptoms or requires active intervention or requires interruption or discontinuation of study medication or the abnormality or investigational value is clinically significant in the opinion of the investigator.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (median treatment duration was 811.0 days, minimum of 43 days and maximum of 1067 days)
Population: Participants in the SAF were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg
Number analyzed (Participants) | 2 | 3 | 3 | 1
Participants | 2 | 3 | 3 | 1

2. Primary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Status at End Of Treattment Visit (EOT)
Description: ECOG performance status was used to assess participants disease progression, and ability to carry out the daily living activities. The participants were graded on a scale of 0 to 5 where 0 = fully active, able to carry on all predisease performance without restriction; 1 = restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 = ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 = capable of only limited self-care,confined to bed or chair more than 50% of waking hours; 4 = completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5 = Dead. Number of participants with ECOG performance status was reported.
Time Frame: EOT Visit (30 days post-last dose, maximum treatement duration of 1067 days)
Population: Participants in the SAF with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg
Number analyzed (Participants) | 2 | 3 | 1 | 1
Participants
  Grade 0 | 2 | 0 | 0 | 0
  Grade 1 | 0 | 3 | 0 | 1
  Grade 2 | 0 | 0 | 1 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (median treatment duration was 811.0 days, minimum of 43 days and maximum of 1067 days)
Arm/Group | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/3 | 2/3 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilteritinib 40 mg (N=2) | Gilteritinib 80 mg (N=3) | Gilteritinib 120 mg (N=3) | Gilteritinib 200 mg (N=1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilteritinib 40 mg (N=2) | Gilteritinib 80 mg (N=3) | Gilteritinib 120 mg (N=3) | Gilteritinib 200 mg (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accommodation disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trichiasis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (5) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Oral mucosal hypertrophy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (5) | 1 (1)
Chronic graft versus host disease in eye (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chronic graft versus host disease oral (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (3) | 0 (0) | 1 (2) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (3) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood insulin abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 1 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lentigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement."

DOCUMENTS (2):
  • Study Protocol (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT02561455/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT02561455/SAP_001.pdf